CLINICAL TRIAL: NCT04584073
Title: Comparison Between the Fate of Secretory Otitis Media in Patients With Adenoids Hypertrophy Undergoing Adenoidectomy Alone or With Myringotomy or With Myringotomy and Tympanostomy Tube Application
Brief Title: Secretory Otitis Media in Adenoids Hypertrophy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Ayman Ahmed Mostafa Abokrisha, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OME in adenoids hypertrophy
Record Dates: First submitted 2020-09-26; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Otitis Media With Effusion
MeSH Terms: conditions — Otitis Media with Effusion | interventions — Adenoidectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adenoidectomy (Active Comparator): Adenoidectomy
  Interventions: Procedure: Adenoidectomy alone or with Myringotomy or with Myringotomy and Tympanostomy Tube application
- Adenoidectomy and Myringotomy (Active Comparator): Adenoidectomy and Myringotomy
  Interventions: Procedure: Adenoidectomy alone or with Myringotomy or with Myringotomy and Tympanostomy Tube application
- Adenoidectomy,Myringotomy and Tympanostomy tube application (Active Comparator): Adenoidectomy and Myringotomy and Tympanostomy tube application
  Interventions: Procedure: Adenoidectomy alone or with Myringotomy or with Myringotomy and Tympanostomy Tube application

INTERVENTIONS:
Procedure: Adenoidectomy alone or with Myringotomy or with Myringotomy and Tympanostomy Tube application — Adenoidectomy with or without tonsillectomy when indicated will be performed. simple Myringotomy incision will be done in the antero-inferior quadrant of pars tensa of both tympanic membranes. Middle ear fluids will be aspirated. Tympanostomy tube application will be done.

SUMMARY:
This study aims to compare the fate of Secretory Otitis Media in patients with adenoids hypertrophy undergoing Adenoidectomy alone or with Myringotomy or with Myringotomy and Tympanostomy Tube application

DETAILED DESCRIPTION:
Otitis media with effusion (OME) is one of the most common diseases during childhood . It is defined as collection of non-purulent effusion (mucoid or serous) in the middle ear space without signs of acute infection. It's synomus are serous otitis media, secretory otitis media or glue ear. Adenoid hypertrophy can cause mechanical obstruction of the Eustachian tube which plays an important role in the pathogenesis of OME.

Management of OME consisted of many varieties; 1- Auto inflation, 2- Medical treatment and 3- Surgical. Surgical treatment indicated in cases where the effusion does not resolve spontaneously or failed medical treatment for 3 months and the main purpose of surgery is to restore middle ear aeration. Treatment options are Adenoidectomy with or without Myringotomy or Myringotomy and Tympanostomy tube application.

The aim of this study is to compare the efficacy of each surgical option in management of otitis media with effusion. This study will be carried out in ENT department of Assiut university hospital on 150 child diagnosed as persistent otitis media with effusion due to adenoid enlargement and they will be categorized randomly into three groups (50 cases per each). Group I will undergo Adenoidectomy alone, group II will undergo Adenoidectomy and Myringotomy and group III will undergo Adenoidectomy and Myringotomy and Tympanostomy tube application. All patients will be subjected to full ENT examination and audiological evaluation. Postoperative evaluation will be done for all patients for 3 months through clinical and audiological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Any case presented with Secretory Otitis Media with adenoids hypertrophy with the following criteria
* Age is between 3 to 17 years old
* With or without chronic tonsillitis
* conductive hearing loss
* Recurrent upper respiratory tract infection
* Dull tympanic membrane on otoscopy (absent cone of light), decreased mobility of tympanic membrane
* Type B tympanogram on tympanometry
* OME not responding to medical treatment for three months

Exclusion Criteria:

* Patients with the following criteria will be excluded from the study
* Previous Myringotomy with or without Tympanostomy Tube application
* Previous adenoidectomy or tonsillectomy
* Previous ear surgery, cleft palate, Down's syndrome, congenital malformation of the ear and cholesteatoma.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Tympanogram | after 3 months of surgery
  Tympanogram is test to measure the movement of tympanic membrane in response to changes in pressure.
Audiogram | After 3 months of surgery
  Audiogram is graph that shows hearing sensitivity

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Popova D, Varbanova S, Popov TM. Comparison between myringotomy and tympanostomy tubes in combination with adenoidectomy in 3-7-year-old children with otitis media with effusion. Int J Pediatr Otorhinolaryngol. 2010 Jul;74(7):777-80. doi: 10.1016/j.ijporl.2010.03.054. PMID 20399511
- [Result] Xu WM, Ye YH. [Effect of tympanostomy tube insertion with adenoidectomy for children with recurrent otitis media with effusion]. Lin Chuang Er Bi Yan Hou Tou Jing Wai Ke Za Zhi. 2016 Dec;30(23):1873-1875. doi: 10.13201/j.issn.1001-1781.2016.23.009. Chinese. PMID 29798016
- [Result] Tian X, Liu Y, Wang M, Liu H. [A systematic review of adenoidectomy in the treatment of otitis media with effusion in children]. Lin Chuang Er Bi Yan Hou Tou Jing Wai Ke Za Zhi. 2014 Apr;29(8):723-5. Chinese. PMID 26248446
- [Result] Hao J, Chen M, Liu B, Yang Y, Liu W, Ma N, Han Y, Liu Q, Ni X, Zhang J. Compare two surgical interventions for otitis media with effusion in young children. Eur Arch Otorhinolaryngol. 2019 Aug;276(8):2125-2131. doi: 10.1007/s00405-019-05421-9. Epub 2019 May 24. PMID 31127413